CLINICAL TRIAL: NCT04427397
Title: The Effects of Using the Sulcular Bristle Tip Technique (SBTT) With an Electric Toothbrush in Reducing Bleeding on Probing and Plaque Removal: A Randomized Control Clinical Trial
Brief Title: Sulcular Bristle Tip Technique (SBTT) With an Electric Toothbrush
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study team has determined that given time and resource restraints, study is to be closed
Sponsor: Tufts University (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Livia Valverde, Assistant Professor, Tufts University School of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00000432
Record Dates: First submitted 2020-06-05; First posted 2020-06-11 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Gum Bleed
Keywords: sulcular bristle tip technique; SBTT; brushing; plaque
MeSH Terms: conditions — Gingival Hemorrhage; Plaque, Amyloid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sulcular Bristle Tip Technique (SBTT) (Experimental): This test group will receive formal instruction on the Sulcular Bristle Tip Technique (SBTT).
  Interventions: Other: Sulcular Bristle Tip Technique (SBTT)
- User manual of the electric toothbrush (DFU) (No Intervention): This control group will be asked to read and use the instructions found in the user manual of the electric toothbrush (DFU). No formal instruction will be provided. The DFU accompany the electric toothbrush regardless of the subject's participation in the research.

INTERVENTIONS:
Other: Sulcular Bristle Tip Technique (SBTT) — Tooth brushing should begin on the distal of the most posterior tooth on one side of the mouth and proceed anteriorly and then posteriorly overlapping areas to the most distal surface of the most posterior tooth on the contra lateral side. The lingual is done in like fashion ending where the brushing began. The opposing arch is brushed in the same manner. When moving from one area to the next, disengage the brush bristles entirely off the teeth to allow them to straighten, and then reposition the brush in the next overlapping area. Do not to drag the bristle tips from one area to the next area. For the lingual of the anterior teeth, the narrow portion of the brush is used with the exact same technique as described above. For the lingual of the mandibular molars, the angulation of the toothbrush bristles to the tooth needs to be somewhat more perpendicular to the tooth than on the buccal to ensure that the bristle tips enter the gingival crevice.
  Arms: Sulcular Bristle Tip Technique (SBTT)

SUMMARY:
In this study, all subjects will be given an electric toothbrush. Half of the participants will be instructed on how to use the Sulcular Bristle Tip Technique (SBTT). The other half of participants will be asked to follow the brushing instructions in the user manual. The study's primary aim is to compare the use of the SBTT with an electric toothbrush in reducing bleeding on probing with the use of an electric toothbrush used without personal professional instruction.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Subjects must show > 20% buccal/lingual cervical sites with bleeding on probing (BoP)
* Subjects must have > 24 natural teeth excluding third molars
* Subjects must have had a professional dental prophylaxis within three months of beginning the study
* Subjects must be willing to brush with electric toothbrush twice daily.
* Subjects who are randomized into Group 1 must be willing to be taught and to demonstrate the SBTT
* Subjects who are randomized into Group 2 must be willing to follow the Sonicare DFU from Philips Oral Healthcare; however, will otherwise be uninstructed until after the study has been completed
* Subjects must be willing to refrain from any oral hygiene for at least 12-18 hours prior to each study follow-up visit.

Exclusion Criteria:

* Subjects who use tobacco products
* Subjects who are currently pregnant (self-reported) due to the greater bleeding tendency caused by hormonal changes
* Subjects with fixed or removable orthodontic appliances
* Subjects whose restorations violate or potentially violate the biologic width.
* Subjects with irregular restoration margins or overhanging margins within 1mm of the crest of the marginal gingiva.
* Antibiotic treatment at the time of the initial examination or during the month prior
* Subjects with cervical probing depth >3 mm
* Subjects with systemic diseases that affect the gingiva
* Subjects taking medications that affect the gingiva
* Subjects who cannot read/write/speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in bleeding on probing (BOP) | Baseline through study completion, an average of 4 months
  To compare the use of the SBTT with an electric toothbrush in reducing BOP with the use of an electric toothbrush used without personal professional instruction.

SECONDARY OUTCOMES:
Effectiveness of professional cleaning | Baseline and 4 months
  To compare whether a dental professional's (DP) cleaning a subject's teeth using an electric toothbrush with the SBTT is more effective in removing cervical plaque than the patient self-cleaning using electric toothbrush with the SBTT at the initial visit and after four months
Change in plaque | Baseline and 4 months
  To compare the plaque removal of each subject at the initial visit with their plaque removal after four months of using the SBTT. To compare the plaque removal of the DP at the initial visit with the DP's plaque removal at the fourth month visit.
Evaluating deformation of toothbrush bristles | Baseline through study completion, an average of 4 months
  To compare the deformation of toothbrush bristles when used by patients using the SBTT with an electric toothbrush with the deformation of the toothbrush bristles with patients using an electric toothbrush uninstructed and whether the deformation is associated with BoP in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Livia Valverde, DMD, Principal Investigator — Tufts University School of Dental Medicine
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States